CLINICAL TRIAL: NCT01158105
Title: Phase 2 Study of Bortezomib (Velcade) for the Treatment of Steroid Refractory Chronic Graft-vs-Host Disease
Brief Title: Bortezomib for the Treatment of Refractory Chronic Graft-vs-Host Disease(cGVHD)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Baylor Research Institute (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 010-037
Record Dates: First submitted 2010-07-06; First posted 2010-07-08 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Graft-versus-host Disease
Keywords: Steroid refractory chronic graft vs host disease (cGVHD); Bortezomib; Velcade
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bortezomib (Experimental): 1.6 mg/m2 intravenous infusion will be administered on days 1, 8, 15, 22 of each 35 day cycle, for up to 6 cycles. Patients who continue to respond during the initial treatment phase with no ongoing significant adverse events will be eligible to receive up to 6 additional cycles. This maintenance dose will be administered on days 1 and 15.
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — 1.6 mg/m2 IV infusion on days 1, 8, 15, 22 of each 35 day cycle, for up to 6 cycles.Patients who continue to respond during the initial treatment phase with no ongoing significant adverse events will be eligible to receive up to 6 additional cycles.This maintenance dose will be administered on days 1 and 15.
  Other Names: Velcade

SUMMARY:
The purpose of this study is to see if bortezomib (Velcade) is effective in the treatment of refractory cGVHD.

DETAILED DESCRIPTION:
Graft vs. host disease represents the most formidable problem following allogeneic hematopoietic stem cell transplantation for hematological diseases. Chronic graft-versus-host disease (cGVHD) is the most serious and common long-term complication of this treatment in patients surviving more than 100 days. Some patients are requiring immunosuppressive therapy for years. cGVHD is associated with a high degree of morbidity and mortality and remains a major cause of late death. When standard treatment with steroids is ineffective or poorly tolerated, effective therapeutic options are limited. Patients with uncontrolled cGVHD with initial therapy including systemic steroids respond poorly to second line options. Recent studies have demonstrated Bortezomib safety in the prophylaxis, and improvement of GVHD suggesting its efficacy.This study is done to evaluate the potential of bortezomib in treating refractory cGVHD.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following inclusion criteria to be enrolled in the study:

* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* ≥18 years old.
* Able to understand and sign informed consent.
* Diagnosis of steroid-refractory cGVHD is defined as either failure to improve after 2 months or progression after 1 month of standard steroid based therapy.
* No previous treatment with Bortezomib for cGVHD
* ECOG PS<3
* Total Bilirubin ≤ 1.5x ULN
* Life expectancy > 3months.
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control for the duration of the study and through a minimum of 30 days after the last dose of bortezomib.
* Male subject agrees to use an acceptable method for contraception for the duration of the study and through a minimum of 30 days after the last dose of study drug.

Exclusion Criteria:

Patients meeting any of the following exclusion criteria are not to be enrolled in the study.

* Patient has a platelet count of <50x 10^9/L within 14 days before enrollment.
* Patient has an absolute neutrophil count of <1.0 x 10^9/L within 14 days before enrollment.
* Patient has a calculated or measured creatinine clearance of <30 mL/minute within 14 days before enrollment.
* Patients with Total Bilirubin > 1.5x ULN
* Patient has ≥ Grade 2 peripheral neuropathy within 14 days before enrollment.
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure (see section 8.4), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
* Patient has hypersensitivity to bortezomib, boron or mannitol.
* Female subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Patient has received other investigational drugs with 14 days before enrollment
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Primary malignancy (for which the transplant was received ) not in remission
* Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.
* Radiation therapy within 3 weeks before randomization. Enrollment of subjects who require concurrent radiotherapy (which must be localized in its field size) should be deferred until the radiotherapy is completed and 3 weeks have elapsed since the last date of therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2010-06; Primary Completion 2013-05 (Actual); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effectiveness and safety of the proteasome inhibitor Bortezomib (Velcade) in the treatment of steroid refractory chronic Graft-vs-Host Disease (cGVHD) | 19 months
  Total time frame including treatment and follow up is 19 months(Maximum of 6 cycles during initial treatment phase, 6 cycles in maintenance phase, and follow up phase for 6 months). Subjects will be assessed for signs and symptoms of cGVHD on day 1 of every cycle using standardized criteria for diagnosis of cGVHD, new clinical scoring system, and new guidelines for global assessment of chronic GVHD severity per NIH consensus development project on criteria for clinical trials in chronic GVHD. Safety will be assessed in terms of adverse events for 30 days following the last dose to a maximum of 6 months. Adverse events will be recorded through out the trial and will be followed by investigator until resolution.

SECONDARY OUTCOMES:
To examine blood cells from patients who develop steroid resistant cGVHD following allogeneic HSCT for disease related gene signatures using DNA microarray analysis techniques | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alan Miller, MD, PhD, Principal Investigator — Charles A. Caner Center, Baylor University Medical Center
Locations (1):
- Charles A. Cancer Center, Baylor University Medical Center, Dallas, Texas, United States